CLINICAL TRIAL: NCT07203612
Title: Prevention of Injuries Among Young Children: Tailoring a Home Supervision Intervention for Latinx Caregivers
Brief Title: Tailoring a Home Supervision Intervention for Latinx Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Michigan University (Other)
Responsible Party: Principal Investigator, Amy Damashek, Principal Investigator, Western Michigan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R15HD097585 (NIH)
Record Dates: First submitted 2025-09-16; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention to increase caregiver supervision and reduce child's risk for injury (Experimental): Group-based intervention to teach caregivers about ways to supervise their children more closely.
  Interventions: Behavioral: SHS
- Control group (Active Comparator): caregivers received information about how to manage common child behavior problems.
  Interventions: Behavioral: Parenting group

INTERVENTIONS:
Behavioral: SHS — Group-based and video-based intervention to teach caregivers of young children how to supervise their children more closely to prevent unintentional injuries.
  Arms: intervention to increase caregiver supervision and reduce child's risk for injury
Behavioral: Parenting group — This intervention was designed to teach caregivers about evidence-based behavioral methods to manage common child behavior problems.
  Arms: Control group

SUMMARY:
The aim of the proposed study is to create and test a modified version of the SHS intervention for Latinx families in Southwest Michigan. We will partner with three nearby Latinx resource centers in addition to a Head Start program that provides preschool to a large number of Latinx families. The project will use an iterative approach to modifying the intervention and will occur in five steps. In step 1, we will conduct focus groups with caregivers and staff from the 3 Latinx resource centers to identify changes to make to the intervention materials. In step 2, we will make modifications to the program materials. In step 3, we will conduct additional focus groups to seek feedback about the revised program materials. In step 4, we will pilot test the revised program materials, and in step 5 we will conduct the RCT of the modified program materials with caregivers of children ages 2-5. We will examine the effect of the modified intervention on caregivers' supervision of their children (using self-reports and observations) and on children's minor injury frequency.

DETAILED DESCRIPTION:
3. APPROACH 3.1 Procedures. The SHS program will be extended to a Latinx population using procedures established by the Centers for Disease Control and Prevention and known as the Map of Adaptation Process. Although there is much diversity within Latinx cultures, the large majority of Latinx families living in Southwest Michigan are of Mexican heritage. Thus, our adaptations will reflect the culture and language of families from Mexico and Central America. The adaptation process emphasizes the need to maintain fidelity of the core elements of an evidence-based intervention like SHS while increasing its relevance (i.e., tailoring it) for a new population. This is achieved by following several steps, which will guide the present study. These steps include: (a) assess the target population's needs (established already by the literature); (b) select an intervention to address those needs (SHS program); (c) prepare the intervention for adaptation (steps 1-3 - see below); and (d) pilot and test the intervention (steps 4-5 below).

Thus, our study will involve an iterative process including five steps. In step 1 we will translate intervention materials (written materials and videos) and conduct focus groups with Latinx caregivers from the community and staff from three Latinx resource centers to identify modifications to be made to program materials. In step 2, the investigators will modify the intervention and video materials based on these focus group data. The investigators anticipate that this step will include making new program videos depicting local Spanish speaking families. The investigators will also make a new introductory video to feature a Spanish speaking narrator. In step 3, the investigators will conduct additional focus groups with Latinx caregivers and center staff using the modified intervention content and make additional changes to the materials if needed. In step 4, the investigators will pilot test the modified intervention with a small group of caregivers and make final modifications. In step 5, the investigators will conduct an RCT to test the modified intervention, including its impact on caregivers' supervision practices and children's injury frequency.

Local Latinx Resource Centers. The investigators will partner with three nearby agencies serving Latinx families: El Concilio (Kalamazoo), Voces (Battle Creek, 30 miles away from campus), and the Hispanic Center of West Michigan (Grand Rapids, 53 miles away). Each agency provides services for Latinx members of their respective communities, including professional translation and interpretation services, liaison services (between families and schools), support regarding immigration and legal issues, assistance accessing resources (e.g., Medicaid, food stamps), youth programs, English as a second language courses, adult education, workforce development and vocational training, and GED classes. Combined, the three Latinx community centers serve approximately 16,000 individuals per year. The Latinx population of each community is as follows: Kalamazoo (5.2%); Battle Creek (7.5%); and Grand Rapids (16.1%; US Census Bureau, 2019).

Head Start. The investigators will also recruit Latinx families from Kent County Head Start. The investigators have successfully collaborated with Kent County Head Start in past research. Head Start is a national program that provides free preschool for l0w-income families of children ages 3-5. The program focuses on kindergarten readiness and also typically provides additional supports for families, such as parental education and linkage to community resources. Kent County Head Start serves approximately 1500 children per year; 30% (450) of these children are Latinx.

Step One: In step 1, the investigators will identify modifications that need to be made to the SHS intervention by conducting 1.5 hour focus groups with both Latinx caregivers of young children (ages 2-5) as well as a focus group with staff from the three Latinx resource centers. Based on recommended sample sizes for focus group research, the investigators will present the SHS materials to Latinx caregivers in three in-person focus groups of 6-8 participants. The investigators will conduct one focus group in each of the Latinx centers from which the investigators will be recruiting (Kalamazoo, Battle Creek, and Grand Rapids). The investigators will conduct one additional focus group including 2-3 agency staff from each of the 3 Latinx serving centers. The investigators will use the SHS materials that have been modified to be appropriate for low-income families from Dr. Damashek's current R15. For these focus groups, the investigators will make preliminary changes to program materials (to make them suitable for the focus group) by translating written materials into Spanish, dubbing video materials to have Spanish voices, and translating subtitles on the videos into Spanish; Morrongiello and her graduate student will make video modifications. Professional translations will be conducted by certified translators at the Latinx resource center in Kalamazoo. Caregiver and staff focus groups will be facilitated by a bilingual RA, in combination with Dr. Damashek. Focus groups will be video recorded and transcribed by a bilingual RA. Transcriptions will be translated into English by a certified translator and will be coded by Drs. Damashek and Morrongiello and URA's to identify themes (i.e., aspects that were helpful about the materials and aspects that need to be changed).

Step 2: Intervention Modification. Themes that emerge from the caregiver and agency staff focus groups will be used to identify modifications that need to be made to the SHS intervention. Dr. Damashek and the bilingual RA's will make new video recordings featuring local Latinx and Spanish speaking families. Families will be recruited from the Latinx resource centers and will be paid $50 for their time (for approximately one hour). The videos will then be edited using equipment available in Dr. Morrongiello's lab to create the final vignettes for the modified program. Dr. Damashek will closely collaborate with Dr. Morrongiello to assist with these edits; they will meet at least biweekly via videochat during this process, as they did in executing the current R15 research together.

Step 3: After changes to the intervention have been made, the investigators will conduct another set of focus groups with Latinx caregivers and agency staff. The investigators will attempt to recruit the same caregivers and staff who attended the original focus groups to determine whether our changes have addressed their concerns and recommendations. If the investigators cannot recruit all the original caregivers and staff, the investigators will recruit additional participants for these focus groups so that the investigators are able to conduct a caregiver focus group of 6-8 participants in each Latinx center as well as a focus group including 2-3 staff from each agency.

Caregiver focus group recruitment and participation. Caregivers will be recruited for the focus groups by distributing information about the focus groups via several approaches. The investigators will provide flyers to be posted in the three Latinx centers, and will also ask them to distribute information about the focus group opportunity via email listserv and social media. The investigators will also distribute flyers for the focus groups via Kent County Head Start. They will distribute flyers to their classrooms and will post them on social media. Materials advertising the focus group opportunity will include text in both Spanish and English and will include a phone number and email for a research staff member who is fluent in Spanish. The research staff will read a recruitment script to the caregiver (in Spanish) and will determine the caregiver's eligibility and interest. Caregivers will be consented at the beginning of the focus group. The investigators will provide focus group participants with $50 gift cards to a local grocery store chain. The investigators will conduct three focus groups (each 1.5 hours in length) with 6-8 caregivers each. In each group, the investigators will explain the purpose of the intervention and show the initial SHS video. Each of the groups will view two (of 6) injury topic video vignettes, so the investigators gain feedback on all six injury topics (falls, drowning, burns, poisoning, choking, guns). Childcare will be provided at the focus groups. The investigators will solicit feedback from agency directors about the days and times that are likely to be most convenient for families to attend the groups, which will be held in person at the Latinx resource centers (one at each center).

Latinx agency staff focus group recruitment and participation. To recruit agency staff for the focus group, the investigators will ask each of the three agency directors to identify several (4-6) staff who would be appropriate to attend the focus group. The investigators will then contact the agency staff via email to provide detailed information about the focus group, and schedule a time to talk to them about their participation via phone or videochat. The staff focus group will be conducted virtually during the regular business day, so that the staff do not have to take personal time to participate in the group. If staff are interested in attending, the investigators will consent them prior to beginning the focus group. Consent will be obtained virtually, via an online data collection tool (Qualtrics), and the investigators will review the consent form with agency staff via phone. The consent form will be provided in Spanish. During the focus group, the investigators will then explain the purpose of the intervention and show them several representative portions of the intervention, including the videos and the problem-solving homework exercises. The investigators will solicit the staff's feedback about the appropriateness of the materials and suggestions for tailoring (e.g., modifications to video vignettes depicting injury-risks at home) to suit their clients. The agency staff will be provided with a $25 gift card for participating.

Both the staff and caregiver focus groups will be audio and video-recorded and transcribed. The transcriptions will then be translated by certified translators at the Latinx resource center in Kalamazoo. Translated transcriptions will be reviewed so that the investigators can identify common suggestions and themes that emerge. The PI Damashek and a bilingual research assistant will facilitate the focus groups, using a structured discussion guide that will be developed in collaboration with Dr. Morrongiello who will observe groups via videochat. The guide will be based on Dr. Morrongiello's prior focus group approach that was used when developing the SHS intervention. Data from these focus groups will then be used to determine additional changes that may need to be made to the intervention materials. Drs. Damashek and Morrongiello will work together to make any additional changes to the intervention.

Step 4: Pilot Test. The investigators will pilot test the modified intervention with one group of 8-10 families and will seek their feedback about the modified intervention materials. The investigators will then make final modifications.

Step 5: RCT. The investigators will use an RCT design to test (N=100 caregivers of children ages 2-5 years) the effects of the modified intervention on caregivers' supervision and children's injury frequency. The control group will not receive any injury prevention intervention, and the treatment group will receive SHS Spanish. The results will be used to support an R01 application to conduct a larger-scale Phase III RCT test of the program.

Graduate and undergraduate research assistants (GRAs and URAs) will play a critical role in all steps of the study. The study will employ one half time GRA at WMU who will be responsible for assisting with recruitment, data collection, and data analysis. The GRA will also be responsible for training and supervising the URAs. The investigators will also hire two bilingual hourly research assistants (RA's) who will assist with study recruitment, facilitate the intervention groups, and conduct data collection. The GRA will accompany the bilingual research staff to assist with data collection and intervention session procedures. Eight undergraduate research assistants (URAs) will assist with the study as well. The URAs will be responsible for data entry, coding of the observations, and providing childcare during data collection and intervention sessions. In addition, a part-time GRA at the University of Guelph (U of G) will assist with preparing video materials, and a Postdoctoral fellow at the U of G will assist with quantitative data analyses.

For the pilot and the RCT, the investigators will use two recruitment methods. The Latinx resource centers will assist in recruiting by sending flyers about the study to their contact lists, posting flyers on their social media pages, providing information about the study at community and in-person meetings, and posting flyers in their buildings. The Grand Rapids resource center will also help to actively advertise the groups by collaborating with the PI to create media interviews (e.g., newspaper). Moreover, this center will share the information with other organizations with whom they partner that serve 2-5 year-olds, including an "Early Learning Neighborhood" that provides early education services to low-income families.

The investigators will also recruit Head Start participants via flyers. Kent County Head Start will distribute study flyers in English and Spanish to individual classrooms as well as via social media and email. The flyers will contain contact information for families to call or email the bilingual RA's. The RA's will call the caregivers and will read a recruitment script. If the caregiver is interested in participating, the RA will give them information about upcoming groups and will sign them up to attend. have been using this recruitment method with Kent County Head Start for the current R15, and it has worked effectively. Caregivers will be eligible to participate if they are the primary caregiver (male or female) for at least one child in the target age range (2-5 years-of-age), if they identify as Latinx, and the caregiver did not participate in the focus group study. The investigators will exclude families in which the target child has been diagnosed with a pervasive developmental disorder or is blind or deaf because such conditions often result in specialized supervision requirements, and the investigators have not tailored the intervention to be appropriate for such families. Later research may examine whether the intervention or a modified version of it, is appropriate for such families. If there is more than one child in the home who is between the ages of 2-5 years, the investigators will use a random procedure to choose the target child. Participants who consent will be randomly assigned to either the treatment or control condition by the primary investigator after the consent appointment.

All data collection and intervention sessions will be conducted in a group format (based on feedback provided by Latinx community center staff). Groups will consist of 8-10 families and will be held at any of the three Latinx resource centers (Kalamazoo, Battle Creek, Grand Rapids). Baseline, post-test, and follow-up assessments will occur during in-person group sessions. Baseline assessments will include three self-report measures of caregiver supervision beliefs and practices, a measure of caregivers' injury beliefs, and a measure of children's injury history. The investigators will also conduct an observational task of caregiver supervision during the group sessions (see description below). All measures have been used in the PI's or Co PI's published research.

The treatment group will participate in four in-person sessions that will include both data collection and delivery of the intervention. The purpose of the combined data collection and intervention delivery is to minimize the amount of response effort required by families and to minimize the likelihood of participant attrition. Moreover, based on feedback from the Latinx resource center directors, the number of intervention sessions has been reduced from 5 (used in the current R15 with low-income families) to 3 sessions to make it more likely that caregivers will attend all sessions (the 4th session is data collection only). At baseline, families in the treatment group will participate in a 2 hour group session; they will complete baseline measures for the first hour of the session and will participate in the first intervention session during the second half of the first session. The second meeting will occur one week later and will only include intervention content. This session will last for 1.5 hours. One week later, participants will attend another 2 hour session, which will include one hour of intervention material (during the first hour) and then one hour of post-test data collection (during the second hour of the group). Participants will then return four weeks later to complete follow-up data collection, which will last for one hour. The control group will participate in three data collection sessions (baseline, post-test, follow-up) that will last for 1 hour each and will follow the same time sequence as the data collection for the treatment group. The post-test session will occur two weeks after baseline, and the follow-up session will occur 4 weeks after the post-test session. The 1-month follow-up will be used to assess for sustainability of effects during which the investigators will administer the same supervision and injury measures as at baseline.

Sessions will be held during convenient hours for families and will include food as well as childcare. If needed, the bilingual RA will assist caregivers with low literacy to complete the measures by reading the measures aloud or by answering questions about the measures. The investigators have used this approach successfully in the current R15. The RA's who deliver the intervention will be trained by Dr. Damashek to deliver SHS and will use a manual to guide delivery (based on previous work, Morrongiello et al., 2017).

The investigators will also collect data on children's minor everyday injury frequencies using a structured injury interview that will be administered weekly via telephone by bilingual RAs; this measure has been used in previous research (including the current R15) by the PI (Damashek & Corlis, 2017). The first interview will be administered in person during the baseline data collection session. Additional administrations will occur weekly via telephone through the follow-up data collection appointment. Caregivers will be paid $40 for each in-person data collection or intervention session and $5 for each phone interview they complete, regardless of the number of injuries reported. Total participation time in the study will be 7 weeks.

3.2 Power Analysis. Effect sizes for the RCT were estimated based on Morrongiello's RCTs testing the SHS and fell within the 'moderate' to 'large' range according to Cohen (1992): ƞ2=.36 for self-report supervision indices, ƞ2=.59 for beliefs, ƞ2=.75 for observational supervision scores. With power set at .80 and p = .05, a sample size of 50 per group (n = 50) will detect a medium to large effect. Thus, a total sample size of 100 will provide sufficient power to detect changes in beliefs and actual supervision. The investigators will recruit participants for the RCT for a period of 2 years. The Head Start program from which the investigators will recruit serves 675 Latinx families over a 2-year period, and the three Latinx resource centers collectively serve 16,000 individuals per year, with an estimated 960 children ages 2-5. This would result in a potential referral base of approximately 1,635. In our current R15, the investigators consented 8% of families into our study. With a potential referral base of 1635 families, the investigators estimate a referral rate of 8%, resulting in 130 participants over a 2-year period. Based on our current R15, the investigators estimate an attrition rate of 15%, leaving a total sample size of 110, which is adequate for our needs.

3.3 Intervention Delivery and Fidelity Assessment. The tailored program will use a detailed manual (modified for group facilitation) to guide delivery of the program and ensure consistency in delivery across participants. The Manual provides week-by-week specification of the materials to use, what is to be covered, questions to be asked, and discussion topics to pursue. It also outlines potential challenges that may arise and provides suggested solutions. Dr. Damashek has been trained by Dr. Morrongiello to implement the intervention, and Dr. Morrongiello will continue to play an active role in program delivery. Dr. Damashek will train the GRA and bilingual RAs to implement the intervention. Each intervention session will be audio recorded. Certified translators will translate and transcribe 20% of sessions (randomly chosen) so that Dr. Damashek can assess fidelity in program delivery. The investigators will use a checklist that the investigators have developed for the current R15, based on the manual, to code fidelity (i.e., coverage of core components). Fidelity checks will be implemented weekly, and Dr. Damashek will meet with the research assistants weekly to provide supervision and discuss any fidelity that may arise.

ELIGIBILITY:
Inclusion Criteria:

* Spanish speaking caregiver of child ages 15 months to 5 years old.

Exclusion Criteria:

* child of caregiver has pervasive develomental disorder, is blink, or deaf.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Supervision Behavior | baseline, immediate post-intervention, 1 month post-intervention
  Caregivers will complete the Computerized Supervision Observation Measure (CSOM), which is a 20-minute observational measure of supervision that was created by Dr. Morrongiello (Morrongiello et al., 2010). The measure assesses the frequency with which caregivers verbally intervene to address risky child behavior (e.g., climbing on a dresser) as well as the type of verbal comment that they make (e.g., prohibitions, directives, or teaching comments). Each parent will view a videotape of a young child (same sex as their own) in a naturalistic home setting. The video will show a child moving throughout the home playing in different areas (living room, kitchen). Parent responses will be coded to rate the degree to which they respond effectively to children' engagement in risky behavior. Coding categories include: prohibitions or threats (e.g., don't do that"), directions or control statements (e.g., "you can put that over there") and teaching/explanations (e.g., "that's hot).
Parent Supervision Attributes Profile Questionnaire (PSAPQ) | baseline, immediately post-intervention, 1 month post intervention
  The PSAPQ will be administered at baseline, immediately post-intervention, and at 1 month post-intervention. The PSAPQ is a measure of parents' supervision practices and beliefs (Morrongiello & Corbett, 2006; Morrongiello & House, 2004). It is comprised of 29 items organized into 4 subscales (protectiveness, supervision, tolerance for risk taking, and belief that fate determines a child's injury risk). Caregivers use a 5-point Likert scale (1= strongly disagree, 5 = strongly agree) to rate the extent to which they agree with items assessing their supervision attitudes and behaviors (e.g., I let my child take some chances in what he/she does; I have my child within reach at all times). The minimum score on the scale is 29, and the maximum score is 145. Higher scores indicate engagement in higher levels of supervision and greater beliefs about the importance of protecting children from injuries.

SECONDARY OUTCOMES:
Injury Frequency Interview | baseline, immediately post-intervention, 1 month post-intervention
  The Injury Frequency Interview is a a structured interview that will be used to assess children' frequency of unintentional injuries throughout the study. An injury will be defined as any unintentional event that caused a physical injury that could be seen (e.g., bruise) or felt (e.g., sprain) by the child or caregiver for a minimum of 1 hour (cf. Morrongiello et al., 2004a). The interviews will be conducted during 5-minute weekly telephone calls that will be completed with caregivers who are enrolled in the study. Weekly reporting is appropriate because minor injuries are difficult to recall over a longer time period (Cummings et al., 2005). Caregivers will be provided with an injury recording sheet to assist with recall during the phone interviews. This study will assess minor injuries because medically attended injuries are a low base rate phenomena and research supports the validity of minor injury assessments as a proxy of more severe or medically attended injuries (Karazsia et a

CONTACTS AND LOCATIONS:
Overall Officials: Amy Damashek, Ph.D., Principal Investigator — Western Michigan University
Locations (1):
- Western Michigan University, Kalamazoo, Michigan, United States

IPD SHARING:
Plan to Share IPD: No